CLINICAL TRIAL: NCT01050309
Title: An Open-label, Single-dose, Three Period Study to Determine the Pharmacokinetic Parameters of Hexaminolevulinate (HAL) Hydrochloride After Vaginal, Enema and Intravenous Administration of Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Berit Nicolaisen/Project Director, Photocure ASA
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: PC CO102/09
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — 5-aminolevulinic acid hexyl ester

ARMS (3):
- Cervix (Active Comparator)
  Interventions: Drug: hexaminolevulinate (HAL)
- colon (Active Comparator)
  Interventions: Drug: hexaminolevulinate (HAL)
- Intravenous (Active Comparator)
  Interventions: Drug: hexaminolevulinate (HAL)

INTERVENTIONS:
Drug: hexaminolevulinate (HAL) — Intravenous dose of HAL 0.4 mg/kg including 100 nCi (3.7 kBq) 14C infused over a one hour period. A vaginal dose HAL 150 mg including 13,9 kBq of 14C HAL will be administered for 7 hours. Following a colon cleaning, 100mg HAL enema including 14,8 kBq of 14C will be instilled for 30 minutes in colon

SUMMARY:
The study will determine the extent of systemic absorption of HAL following vaginal and enema administration compared to intravenous administration to healthy female volunteers.

In addition, the pharmacokinetic parameters for the combined level of 14C labelled substances (sum of parent and possible metabolites)will be assessed. The safety and tolerability of HAL following vaginal, enema and intravenous administration to healthy female volunteers will be investigated.

DETAILED DESCRIPTION:
This is a single-centre, non-randomised, open-label, single-dose, three-period study planned to include eight healthy female volunteers. Subjects will attend a screening visit within 21 days of dosing. In Period 1, an intravenous dose of HAL 0.4 mg/kg including 100 nCi (3.7 kBq) 14C will be infused over a one hour period. In Period 2, a vaginal dose HAL 150 mg including 13,9 kBq of 14C HAL will be administered for 7 hours. In period 3, following a colon cleaning, 100mg HAL enema including 14,8 kBq of 14C will be instilled for 30 minutes in 8 subjects. Period 1, 2 and Period 3 will be conducted in an identical manner except that subjects will receive the HAL by different dose routes. Blood samples will be drawn during 3 days of follow up to evaluate the single dose pharmacokinetics of HAL for each dose route. In addition, urine and faeces will be collected from Period 1. The urine and faces samples will be stored for possible future analysis.

There will be a minimum of 7 days washout between the three dosing periods. Subjects will attend a final follow-up visit at the 14 day blood sampling visit in the third study period. The total amount of 14C-label used in each volunteer is estimated to be approximately 33.3 kBq. No formal calculation of the radiation burden was made. Based on data of full-dose ADME studies it is estimated that this dose will give a radiation burden of less than 0.01 mSv, which falls in ICRP category I: trivial risk.

Diagnosis and main criteria for inclusion:

Healthy female subjects aged 18 to 55 years (inclusive) with body mass index (BMI) >19 and <30 kg/m2 who give written informed consent and comply with all the inclusion and exclusion criteria, will be entered into the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy women aged 18 to 55 years (inclusive)
* Body Mass Index (BMI) > 19 and < 30 kg/m2
* Able to understand the nature of the study and to give written informed consent

Exclusion Criteria:

* consumption of medication (including 'over the counter' preparations and herbal remedies) within two weeks of dosing. Simple analgesics (e.g. paracetamol) may be allowed at the discretion of the Investigator
* past or current drug exposure amounting to drug abuse or addiction
* past or current alcohol exposure amounting to alcohol abuse or addiction; [i.e. > 21 units per week for females, where 1 unit = one measure of spirit (25 ml), one glass of wine (125 ml) or ½ pint beer]
* smokers of more than five cigarettes a day
* donation of blood within two months before the study
* receipt of a 14C labelled compound in one year before the study
* participation in a clinical trial involving receipt of a licensed or unlicensed medicinal product within three months before the study
* unwilling or unable to comply with the study protocol for any reason
* positive test for hepatitis B surface antigen or hepatitis C antibody or human immunodeficiency virus (HIV) at screening
* subjects with childbearing potential (i.e. pre-menopausal, not surgically sterile) not willing to use a medically accepted contraceptive (oral contraception) regimen from the pre-study screening until at least 3 months after the last study period.
* pregnant or lactating women
* clinically relevant abnormalities in the pre-study screening.
* known allergy or intolerance to any compound in the test product or any other closely related compound
* any other acute or chronic disease which could influence the subject's health and/or the study results, e.g. porphyria
* clinically relevant abnormalities from standard gynecological examination (incl. cervical smear and determination of position of uterus)
* Irregular defecation pattern, i.e. less than once per 2 days

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the extent of systemic absorption of HAL following vaginal and enema administration compared to intravenous administration to healthy female volunteers.

SECONDARY OUTCOMES:
To determine pharmacokinetic parameters for the combined level of 14C labelled substances. To assess the safety and tolerability of HAL following vaginal, enema and intravenous administration to healthy female volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Berit Nicolaisen, M.Sc., Study Director — Photocure ASA
Locations (1):
- Pra-Eds-Nl, Zuidlaren, Netherlands